CLINICAL TRIAL: NCT00930592
Title: Assessor-Blinded Study of the Metabolic Syndrome and Surrogate Markers of Increased Cardiovascular Risk in Children With Moderate to Severe Psoriasis Compared With Age Matched Population of Children With Warts
Brief Title: Peds Metabolic Syndrome in Psoriasis
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: Peds Metabolic Syndrome
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis; Metabolic Syndrome
Keywords: Psoriasis; Metabolic Syndrome; Cardiovascular Risk
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with Psoriasis: Children and adolescents from 10-17 years of age with moderate to severe psoriasis.
- Control: children with warts: Children and adolescents from 10-17 years of age with warts.

SUMMARY:
The objective of this study is to assess whether there is an increased risk of the metabolic syndrome in children with psoriasis compared to children without psoriasis.

DETAILED DESCRIPTION:
Adult patients with psoriasis, especially those who are young and with severe disease, have an increased prevalence of myocardial infarction and metabolic syndrome, and increased mortality. Tumor Necrosis Factor (TNF) and other inflammatory cytokines are felt to play an important role not only in the pathogenesis of psoriasis and psoriatic arthritis, but in the pathogenesis of the metabolic syndrome and increased cardiovascular mortality and morbidity.

However, the prevalence of metabolic syndrome and surrogate markers of increased cardiovascular risk, such as lower flow-mediated dilation (FMD) during reactive hyperemia, measured by high-resolution brachial artery ultrasound, lower hyperemia-induced, pulse wave amplitudes as measured by finger plethysmograph peripheral artery tonometry, and elevated blood CRP levels, in children with psoriasis, are unknown.

We will use the definition of metabolic syndrome described by de Ferranti: Participants are defined as having metabolic syndrome if they meet or exceed the criteria for 3 or more of the following 5 variables: 1) triglycerides ≥1.1 mmol/L; 2) HDL cholesterol <1.3 mmol/L; 3) fasting blood glucose ≥6.1 mmol/L; 4) waist circumference (cm) >75th percentile for age and sex; and 5) systolic or diastolic blood pressure (mm Hg) >90th percentile for age, sex, and height.

The following two noninvasive procedures will be used to assess additional cardiovascular risk: flow mediated dilation (FMD) and finger plethysmography peripheral artery tonometry (PAT). These procedures have been used extensively to measure adults for clinical study purposes for many years.

As a control group, we will compare children with psoriasis to age-, race-,and gender-matched children with warts.

ELIGIBILITY:
Inclusion Criteria:

* 10-17 year old children with either moderate to severe psoriasis or with warts
* For psoriasis patients, body surface area covered must be 5% or more or must have had a documented history of 5% or more body surface area involvement
* Ability to understand and sign an age-appropriate consent form
* Parent or Guardian over 18 years old able to understand and sign consent form

Exclusion Criteria:

* Psoriasis or wart patient younger than 10 or 18 years or older
* For psoriasis patients, body surface area covered less than 5% or have not had a documented history of 5% or more body surface area involvement
* Inability of child or adult parent/guardian to understand or sign consent
* Pregnant or lactating females.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: These subjects will be recruited from the pediatric Dermatology Clinic at Tufts Medical Center, community physician referral, and advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine if children with psoriasis will have an increased prevalence of the metabolic syndrome. | one assessment

SECONDARY OUTCOMES:
Metabolic syndrome in children with psoriasis will be determined using body weight, BMI, waist circumference, blood pressure, fasting blood sugar, and blood lipid profile. | one assessment
Surrogate endpoints indicating potential increased cardiovascular risks, including high sensitivity CRP, flow-mediated dilation (FMD) during reactive hyperemia, and hyperemia-induced, pulse wave amplitudes. | one assessment
For psoriasis patients only: PASI, BSA, and PGA will be measured to establish extent of disease. | one assessment
Safety Outcome Measures: All adverse events (AEs) will be recorded and monitored. | each occurance

CONTACTS AND LOCATIONS:
Overall Officials: Alice B. Gottlieb, M.D., PhD., Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelfand JM, Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006 Oct 11;296(14):1735-41. doi: 10.1001/jama.296.14.1735. PMID 17032986
- [Background] Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB, Gelfand JM. Prevalence of cardiovascular risk factors in patients with psoriasis. J Am Acad Dermatol. 2006 Nov;55(5):829-35. doi: 10.1016/j.jaad.2006.08.040. Epub 2006 Sep 25. PMID 17052489
- [Background] Gottlieb AB, Dann F, Menter A. Psoriasis and the metabolic syndrome. J Drugs Dermatol. 2008 Jun;7(6):563-72. PMID 18561588
- [Background] Huang PH, Chen JW, Lu TM, Yu-An Ding P, Lin SJ. Combined use of endothelial function assessed by brachial ultrasound and high-sensitive C-reactive protein in predicting cardiovascular events. Clin Cardiol. 2007 Mar;30(3):135-40. doi: 10.1002/clc.20058. PMID 17385705
- [Background] Strober B, Teller C, Yamauchi P, Miller JL, Hooper M, Yang YC, Dann F. Effects of etanercept on C-reactive protein levels in psoriasis and psoriatic arthritis. Br J Dermatol. 2008 Aug;159(2):322-30. doi: 10.1111/j.1365-2133.2008.08628.x. Epub 2008 May 22. PMID 18503600
- [Background] Shapiro J, Cohen AD, David M, Hodak E, Chodik G, Viner A, Kremer E, Heymann A. The association between psoriasis, diabetes mellitus, and atherosclerosis in Israel: a case-control study. J Am Acad Dermatol. 2007 Apr;56(4):629-34. doi: 10.1016/j.jaad.2006.09.017. Epub 2006 Dec 8. PMID 17157411
- [Background] Paller AS, Siegfried EC, Langley RG, Gottlieb AB, Pariser D, Landells I, Hebert AA, Eichenfield LF, Patel V, Creamer K, Jahreis A; Etanercept Pediatric Psoriasis Study Group. Etanercept treatment for children and adolescents with plaque psoriasis. N Engl J Med. 2008 Jan 17;358(3):241-51. doi: 10.1056/NEJMoa066886. PMID 18199863
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Rand WM, Udelson JE, Karas RH. Peripheral vascular endothelial function testing as a noninvasive indicator of coronary artery disease. J Am Coll Cardiol. 2001 Dec;38(7):1843-9. doi: 10.1016/s0735-1097(01)01657-6. PMID 11738283
- [Background] Haller MJ, Stein J, Shuster J, Theriaque D, Silverstein J, Schatz DA, Earing MG, Lerman A, Mahmud FH. Peripheral artery tonometry demonstrates altered endothelial function in children with type 1 diabetes. Pediatr Diabetes. 2007 Aug;8(4):193-8. doi: 10.1111/j.1399-5448.2007.00246.x. PMID 17659060
- [Background] de Ferranti SD, Gauvreau K, Ludwig DS, Neufeld EJ, Newburger JW, Rifai N. Prevalence of the metabolic syndrome in American adolescents: findings from the Third National Health and Nutrition Examination Survey. Circulation. 2004 Oct 19;110(16):2494-7. doi: 10.1161/01.CIR.0000145117.40114.C7. Epub 2004 Oct 11. PMID 15477412